CLINICAL TRIAL: NCT06469489
Title: Safety and Adequacy of Trans-jugular Liver Biopsy in Patients With Liver Disease: SAFE-TJLB Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-SAFE-TJLB
Record Dates: First submitted 2024-01-03; First posted 2024-06-21 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Disease patients undergoing Trans-Jugular Liver Biopsy
  Interventions: Other: Liver Disease of all etiologies

INTERVENTIONS:
Other: Liver Disease of all etiologies — No intervention

SUMMARY:
Liver biopsy is considered the gold standard for the evaluation of acute and chronic liver disorders. Liver biopsy provides information regarding diagnosis, disease progression, and response to therapy in patients with chronic liver diseases. Trans-jugular liver biopsy (TJLB) consists of obtaining liver tissue through a rigid cannula introduced into one of the hepatic veins typically using jugular venous access. This approach reduces the risk of hemorrhage after biopsy because the bleeding resulting from the biopsy needle will drain into the hepatic veins. In the past, the specimens obtained by a transjugular approach were considered suboptimal compared with the samples obtained with percutaneous needles because they were smaller and more fragmented. TJLB was initially indicated for patients who had a contraindication to percutaneous biopsy such as those with a coagulopathy or congenital clotting disorders, ascites, acute liver failure, large amount of adipose tissue, and patients after liver transplantation. The clinical role of TJLB has expanded due to the possibility of performing hemodynamic evaluation of the hepatic and portal venous systems, which provides useful information and may guide therapy in patients with portal hypertension.

Lacuna in literature:

There is no prospective study in India evaluating the safety and efficacy of trans-jugular liver biopsy in patients with liver disease.

DETAILED DESCRIPTION:
Hypothesis:

Trans-jugular liver biopsy is safe, gives adequate sample for pathological examination in patients with liver disease.

Aim of study:

To evaluate safety and adequacy of trans-jugular liver biopsy in patient with liver disease.

Primary objective:

1. Adequacy of trans-jugular liver biopsy
2. Safety of trans-jugular liver biopsy

Secondary objective:

1. Indications of liver biopsy
2. Procedural time (in and out of catheter)
3. Number of passes
4. Failure rate
5. Day care time
6. VAS: pain (Abdomen and Neck, pre and post procedure)
7. Complications- arrythmia, hematoma
8. Time of Fluro exposure

Patients and methods Study Design A prospective, observational cohort study will be conducted in patients with suspected or known liver disease between November 2023 to May 2024 at the Institute of Liver and Biliary Sciences (ILBS), New Delhi.

Clinical protocol An informed consent was taken from patients with liver disease undergoing liver biopsy as per clinical indication. The following demographic data was recorded at inclusion: Age, gender, co-morbidities, type, and etiology of liver disease. Laboratory parameters include complete blood count, liver function tests, kidney function tests, INR. Severity of liver disease (MELD score, CTP score, AARC score).

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years age.
2. Patient with suspected or known liver disease undergoing trans-jugular liver biopsy as per clinical indication.

Exclusion Criteria:

- None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver Diseases of all etiologies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with liver biopsy taken of more than 1.5 cm in length | Day 0
Adverse event | Day 7

SECONDARY OUTCOMES:
Procedural time (in and out of catheter) | Day 0
Number of passes | Day 0
Failure rate | Day 0
Day care time | Day 1
VAS: pain (Abdomen and Neck, pre and post procedure) | Day 0
  VAS=10 is maximum pain
Number of patients with Complications- arrythmia, hematoma | Day 0
Time of Fluro exposure | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided